CLINICAL TRIAL: NCT02748876
Title: A Randomised Cross-over Pilot Study of the Effect of His-Ventricular (HV) Interval Optimisation in Cardiac Resynchronisation Therapy
Brief Title: Effect of His-Ventricular (HV) Interval Optimisation in Cardiac Resynchronisation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- His-Ventricular (HV)-optimised (Experimental): His-Ventricular (HV) optimised atrioventricular delay
  Interventions: Other: His-Ventricular (HV) optimisation
- Non-optimised (No Intervention): Standard atrioventricular delay

INTERVENTIONS:
Other: His-Ventricular (HV) optimisation — Optimisation of atrioventricular pacing interval
  Arms: His-Ventricular (HV)-optimised

SUMMARY:
Cardiac resynchronisation therapy (CRT) is a specialised type of pacemaker used in patients with severe heart failure to improve symptoms and survival. Approximately one third of patients treated with CRT do not notice significant improvement in their symptoms and this may be due to inadequate co-ordination between the upper and lower chambers of the heart (atrioventricular dyssynchrony).

The investigators propose a new method to achieve atrioventricular synchrony in CRT based on measurements of electrical conduction from within the heart. Patients referred for CRT implantation at Castle Hill Hospital are eligible to participate. During CRT implantation, additional measurements, will be recorded from within the heart. After implantation, device settings will be adjusted to either standard or electrophysiologically-optimised settings with cross-over at 4 months.

The investigators hypothesis is that patients with optimised settings will derive additional benefit compared to patients with standard pacemaker-determined settings.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure
* Referred for cardiac resynchronisation therapy (CRT) with or without defibrillator
* In sinus rhythm
* Patients must have a telephone
* Ability to give informed consent
* Ability to complete the study

Exclusion Criteria:

* Severe valve disease or previous valve replacement
* Previous atrial flutter ablation
* Chronic kidney disease Stage 3 or above
* Recent myocardial infarction
* Ongoing cardiac ischaemia
* Infiltrative cardiomyopathy
* Wolff-Parkinson White syndrome
* Presence of second or third degree heart block
* <90% biventricular pacing at 3 months
* Hypertrophic cardiomyopathy
* Pregnancy or breastfeeding
* On treatment for hypothyroidism or hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Change in amino-terminal pro-B-type natriuretic peptide (NT-proBNP) | 7 months and 11 months

SECONDARY OUTCOMES:
Increase in 6-min walk test distance by ≥25 m | 7 months and 11 months
≥5points improvement in the short Kansas City Cardiomyopathy Questionnaire score | 7 months and 11 months
Reduction of left ventricular end-diastolic volume. | 7 months and 11 months

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No